CLINICAL TRIAL: NCT02028468
Title: Anterolateral Watson Jones Approach Versus Transgluteal Approach for Uncemented Hemi- Arthroplasty in Displaced Femoral Neck Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 811419
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2022-03

CONDITIONS: Femoral Neck Fracture
Keywords: Femoral Neck Fracture; Anterolateral approach; Trans-gluteal approach; Watson Jones approach; Hardinge approach
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Hemiarthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Anterolateral Approach (Active Comparator): Patient Operated with Watson Jones Approach
  Interventions: Procedure: hemiarthroplasty
- Trans-gluteal Approach (Active Comparator): Patient operated with Trans-gluteal Hardinge Approach
  Interventions: Procedure: hemiarthroplasty

INTERVENTIONS:
Procedure: hemiarthroplasty

SUMMARY:
Hemiarthroplasty is a well established treatment of Femoral Neck Fractures in the Elderly. During the last decade the use of Minimal Invasive Surgical( MIS) approaches have been increasing. Our hypothesis is that Patients with a Femoral Neck Fracture may benefit from a MIS approach.

DETAILED DESCRIPTION:
The study's main objective: The purpose of the study is to test the following hypothesis. Patients 70 to 90 years with a displaced femoral neck fracture, operated with a hemiarthroplasty through an anterolateral approach, have less pain and better patient satisfaction as measured by PROMs than patients operated through the lateral approach.

The study's subsidiary objectives. We aim to shed light on the following subsidiary hypotheses.

1. A hemiarthroplasty inserted through an anterolateral approach gives less bone resorption, as measured by DEXA around the stem, than a hemiarthroplasty inserted via a direct lateral approach.
2. A hemiarthroplasty inserted through an anterolateral approach causes lesser degree of muscle damage, as measured by CK, than a direct lateral approach

ELIGIBILITY:
Inclusion Criteria: Patients 70- 85 Years of Age -

Exclusion Criteria:

Dementia, Infection Not Suitable for Hemiarthroplasty

-

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-03 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale Pain and Patient Satisfaction | Pre and postoperative, 3 and 12 Months

SECONDARY OUTCOMES:
Timed up and go | postoperative, 3 and 12 Monthes
  TUG test- Timed up and Go
Harris Hip Score | Pre / Postoperative, 3 and 12 Months
Hip Osteoarthritis Disability Score | Postoperative, 3 and 12 Months
EuroQol | Postoperative, 3 and 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, Professor, Principal Investigator — University of Oslo Ullevål
Locations (1):
- Sorlandet Hospital, Kristiansand, Norway

REFERENCES:
- [Derived] Ugland TO, Haugeberg G, Svenningsen S, Ugland SH, Berg OH, Pripp AH, Nordsletten L. Biomarkers of muscle damage increased in anterolateral compared to direct lateral approach to the hip in hemiarthroplasty: no correlation with clinical outcome : Short-term analysis of secondary outcomes from a randomized clinical trial in patients with a displaced femoral neck fracture. Osteoporos Int. 2018 Aug;29(8):1853-1860. doi: 10.1007/s00198-018-4557-y. Epub 2018 May 22. PMID 29789919